Consent for children 14-17 years old

**Title of Research Study:** Promote Healthy Lifestyle Behaviors for Adolescents with Mental Health Conditions

**Principal Investigator:** Rachel Sharp, BSN, RN, CPN, DNP-FNP Student, Florida State University College of Nursing

*Faculty Advisor*: Dr. Geneva Scott-King, DNP-MSN-FNP-C, Teaching Faculty II, Florida State University College of Nursing

## What is this study about?

A study is usually done to understand how things work or to find a better way to take care of people. You are being asked to take part in this research study because you are an adolescent, 14-17 years old, currently diagnosed with a mental health condition(s)

# What should I know about a research study?

In this study, I want to find out more about the impact of an educational intervention on improving healthy lifestyle knowledge and behaviors (nutrition, physical activity, screen time, and sleep). You do not have to be in this study if you do not want to do so. It is up to you if you want to take part. You can choose not to take part now and change your mind later if you want. Your decision will not be held against you. You can ask all the questions you want before you decide.

### How long will the research last?

• I expect that you will be in this research study for one- month. Within a two-week period, you will be asked to complete a pre-survey questionnaire that takes approximately 10-15 minutes and attend an online Zoom educational session that takes approximately 45 minutes. One-month after completing the pre-survey and educational session, you will be asked to take a post-survey questionnaire that will take approximately 10-15 minutes.

# What happens if I say "Yes, I want to be in this research"?

If you agree to be in this study, you will be asked to answer questions and join an online educational session with your parent(s)/legal guardian(s) on healthy lifestyle knowledge and behaviors

- You will receive a project pre-survey questionnaire via your e-mail in the middle to end of September 2022. You will have 2 weeks to complete pre-survey and attend zoom educational session.
- You will be invited to attend an online Zoom educational session with your parent(s)/legal guardians(s). A reminder email will be sent to you to complete the

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152

survey. The educational session will be recorded and sent via email 1 week after education session.

- You will then receive a post-survey 1 month after and participate in an online educational session in the middle to end of October 2022.
- Study will be completed by early November 2022.

### Is there any way being in this study could be bad for me?

There is nothing bad that will happen to you although there is minimal risk associated with this study. That means you may feel embarrassed with some of the questions that I will ask, or you may feel uncomfortable answering some of my questions. Taking the questionnaires and joining the educational presentation may make you tired. You can skip any questions you do not want to answer/not do something if you don't want to/stop taking part at any time.

## What happens to the information collected for the research?

• We will do everything that we can to protect and secure any information about you that we collect. Your information will only be shared only with people have must review this information. We cannot promise complete secrecy, but we will work to keep your name and other information private.

#### What else do I need to know?

If you agree to take part in this study, the adolescent-parent/legal guardian dyad will receive a \$5.00 Amazon E-Gift Card with completion of the 3 activities associated with the project: presurvey, educational presentation, and post-survey. E-Gift Cards will be sent to email provided via questionnaire (REDCap) for adolescent-parent/legal guardian dyad. You will receive compensation within 24-48hrs after completing each activity of the project. Total compensation for dyad is \$15.00 in Amazon E-Gift Cards when project is completed in its entirety. Withdrawing or discontinuing taking part in the study will preclude participants from earning further incentive

#### Who can I talk to?

If you have any questions or complaints about the study, you can talk to your parents or you can talk to the research team at

Mrs. Rachel Sharp, BSN, RN, CPN
FSU DNP-FNP Student
Florida State University College of Nursing
rls14c@my.fsu.edu

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152

Dr. Geneva Scott-King, DNP-MSN-FNP-C

Teaching Faculty II

Florida State University College of Nursing gscottking@fsu.edu

• You can also talk with the people that reviewed and approved this study. They can be reached at 850-644-7900, or <a href="https://humansubjects@fsu.edu">humansubjects@fsu.edu</a> or Baptist Health IRB at 904-202-2127 or <a href="https://Baptist.IRB@bmcjax.com">Baptist.IRB@bmcjax.com</a>.